CLINICAL TRIAL: NCT01032577
Title: Prospective Study Comparing the Sensed R Wave in Bipolar and Extended Bipolar Configurations
Brief Title: A Study Comparing the Sensed R Wave in Bipolar and Extended Bipolar Configurations
Acronym: PropR
Status: Completed | Type: Observational
Sponsor: Trinity Health Of New England (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-01-005-E
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Ischemic and Nonischemic Cardiomyopathy, With Primary and Secondary Implant Indications
Keywords: ischemic cardiomyopathy; nonischemic cardiomyopathy; implant; bipolar sensing; extended bipolar sensing
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cardiomyopathy, with implant indications: 30-50 volunteers age >18, male and female with ability to give informed consent, who are expected to live more than one year, with indication for defibrillator implant and who are not pacemaker dependent.

SUMMARY:
The PropR study will evaluate sensing during ventricular fibrillation (VF) in both bipolar and extended bipolar configurations, in order to evaluate if both can be used interchangeably in caring for patients. In addition, follow up evaluation of R wave amplitude over time would allow us to determine whether one configuration is more likely to be associated with change. This understanding would be important in selecting the proper configuration at the time of implant.

DETAILED DESCRIPTION:
Hypothesis:

Sensing in bipolar and extended bipolar configurations are the same. However, sensing in bipolar over time is more likely to decrease when compared to extended bipolar.

Objectives:

1. To compare bipolar sensing and extended bipolar sensing in VF.
2. Compare sensing in bipolar and extended bipolar over time.

Methods:

1. This study will be a randomized comparison of bipolar and extended bipolar sensing. As per usual standard of care, at the end of ICD implantation two sensing tests in VF will be performed. Patients will be randomized to sensing in VF through the device. Each patient will undergo testing in one randomized configuration followed by a second test in the other configuration. After testing at the time of implant, each patient will be seen at one month in follow up. Sensing of each configuration will be reevaluated at that time in sinus rhythm.
2. Each patient will serve as their own control, as data for sensing in both configurations will be obtained in VF at the time of implant. During testing both signals types will be recorded simultaneously through the ICD. The primary endpoint will be duration of sensing (time to detection) in VF at the time of implant.
3. The secondary endpoint will be sensing in sinus rhythm at one month.
4. The patient population will include approximately 30-50 volunteers age >18, male and female, both ischemic and nonischemic cardiomyopathy, with primary and secondary implant indications.
5. Patients will be recruited when being evaluated for defibrillator implant.
6. Inclusion criteria: age >18 with ability to give informed consent, who are expected to live more than one year, with indication for defibrillator implant and who are not pacemaker dependent. Patients will have either ischemic or nonischemic cardiomyopathy.
7. Exclusion criteria: age <18, inability to give informed consent, or life expectancy less than one year, pacemaker dependence, or use of preexisting lead for sensing, any condition which would preclude ICD testing at the end of the implant. Patients who are undergoing upgrade to an ICD from a pacemaker will also be excluded. In addition, patients with inherited arrhythmias or ion channel related arrhythmias will be excluded from the study.
8. Withdrawal criteria: inability to implant device, implant lead at the RV apex, or make follow up appointment (living out of state), patient death at time of implant, elevated DFT (<10 J margin between DFT and maximum output of the device) requiring additional procedures, subcutaneous array etc.
9. Duration of patient participation would be one month.
10. Duration of study would be one year.

Procedures:

1. Procedures to be followed would include screening of all eligible patients undergoing implant of a Medtronic defibrillator for either primary or secondary prevention. If patients meet inclusion criteria they would then undergo informed consent and if willing be enrolled in the study. Defibrillator implant and testing would be performed as per usual practice of the implanting physician. The RV lead will be placed at the RV apex as is usual for regular implantation of devices. However, if a lead is placed elsewhere, the patient will need to be withdrawn from the study.
2. When VF induction is performed, sensing configuration would be tested in a randomized fashion, unblinded to the operator. The untested configuration would then be tested during second VF induction. Both tests would be performed at a sensitivity setting of 1.2mV, with a number of intervals to detection (NID) of 24/32. Final programming polarity will be left at the initially tested polarity (first DFT test), unless the operator sees a need to program differently for patient safety reasons.
3. Medtronic defibrillators with both sensing configurations available will be used. Data collection will be performed by Dr. Tolat, Dr. Berns, Dr. Lippman, Dr. Dell'Orfano, and the study coordinator involved with the study. A data collection form and spreadsheet will be kept for use when collecting data for analysis. Follow up will be performed at one month post implant in the office.

Risk Analysis:

1. Anticipated risks are no more than that anticipated with usual ICD implant. To date, usual implant includes induction of VF with analysis of sensing in VF and evaluation of defibrillation threshold by delivery of shock.
2. There is no expected increased exposure to risk by performing this study.
3. Potential benefits would include gathering additional information on sensing in VF in both configurations instead of performing the two sensing tests in one configuration. This may directly benefit the patient by allowing for reprogramming defibrillator without bringing the patient back to the hospital for further testing.

Data Analysis:

1. Data collection will include patient information kept in a database with name kept confidential. Patients will only be identified by number in keeping with privacy laws and practice. In addition to usual patient characteristics, data variables to be collected in both configurations will include: R wave amplitude in sinus rhythm, time to detection in VF, total episode duration (time to Vfib detection and charge delivered), number of "drop outs" (undersensing) in VF, and follow up R wave amplitude in one month.
2. Statistical Methods will compare bipolar sensing configuration to the extended bipolar configuration at baseline, sensing in VF (as measured by "drop out", time to detection), and follow up amplitude of the R wave at one month.
3. The current expected sample size with this pilot study is 30 patients. This may require reevaluation depending on results at the time of interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 with ability to give informed consent,
* patients who are expected to live more than one year,
* patients with indication for defibrillator implant,
* patients who are not pacemaker dependent,
* patients with either ischemic or nonischemic cardiomyopathy.

Exclusion Criteria:

* age < 18,
* inability to give informed consent,
* life expectancy less than one year,
* pacemaker dependence, or use of preexisting lead for sensing,
* any condition which would preclude ICD testing at the end of the implant,
* patients who are undergoing upgrade to an ICD from a pacemaker will also be excluded,
* patients with inherited arrhythmias or ion channel related arrhythmias will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will include approximately 30-50 volunteers age >18, male and female, both ischemic and nonischemic cardiomyopathy, with primary and secondary implant indications.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Duration of sensing (time to detection) in VF at the time of implant. | At implant

SECONDARY OUTCOMES:
Sensing in sinus rhythm at one month | One month post implant

CONTACTS AND LOCATIONS:
Overall Officials: Aneesh Tolat, MD, Principal Investigator — Attending Cardiac Electrophysiologist, St Francis Hospital and Medical Center
Locations (1):
- St Francis Hospital and Medical Center, Hartford, Connecticut, United States